CLINICAL TRIAL: NCT00003176
Title: A Phase II Trial of Temozolomide and BCNU for Anaplastic Gliomas
Brief Title: Temozolomide and Carmustine in Treating Patients With Anaplastic Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NABTC-9701; CDR0000065986 (Registry Identifier: PDQ (Physician Data Query)); NCI-T96-0082
Record Dates: First submitted 1999-11-01; First posted 2004-04-07 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Glioma; Gliosarcoma | interventions — Carmustine; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: carmustine
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of temozolomide and carmustine in treating patients with anaplastic glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the activity, measured in terms of progression free survival, of carmustine plus temozolomide in recurrent glioblastoma. II. Estimate the response rate of recurrent glioblastomas to this combination. III. Estimate the response rate of newly diagnosed anaplastic astrocytomas and mixed anaplastic glioma to this combination. IV. Evaluate the qualitative and quantitative toxicities of this combination in patients with anaplastic gliomas.

OUTLINE: This is a nonrandomized study. Patients are stratified by disease (recurrent glioblastoma vs anaplastic astrocytoma or mixed anaplastic glioma). Patients receive carmustine intravenously on day 1 two hours prior to temozolomide. Temozolomide is administered orally on day 1. Cycles repeat every 42 days. Treatment for patients with recurrent glioblastoma may continue for 8 cycles in the absence of disease progression or unacceptable toxicity. If there is no disease progression after 8 cycles, treatment may continue further at the investigator's discretion. Patients with anaplastic astrocytoma or mixed anaplastic glioma continue for 4 cycles of treatment. Patients are followed periodically at the investigator's discretion, at least twice in the first 4 months, and then until death.

PROJECTED ACCRUAL: A minimum of 17 patients and a maximum of 37 patients will be accrued in the recurrent glioblastoma stratum and 45 patients will be accrued into the anaplastic astrocytoma and mixed anaplastic glioma stratum.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant glioma - Recurrent glioblastoma - Anaplastic astrocytoma - Mixed anaplastic glioma For recurrent glioblastoma: Required documented progression must include an increase in tumor size of at least 25% or appearance of new lesion For anaplastic astrocytoma or mixed anaplastic glioma: Must have measurable, contrast enhancing disease on postoperative CT or MRI scan No postoperative radiation or chemotherapy If patients have received prior brachytherapy or stereotactic radiosurgery, they must have confirmation of true progressive disease rather than radiation necrosis by PET scanning or biopsy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 1,800/mm3 Platelet count at least 125,000/mm3 Hemoglobin at least 9 g/dL (transfusion allowed) Hepatic: Bilirubin less than 1.5 mg/dL SGOT less than 2.0 times upper limit of normal Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 70 mL/min Cardiovascular: No uncontrolled arrhythmias or conduction defects No unstable or newly diagnosed angina pectoris No New York Heart Association class II-IV heart disease No congestive heart failure No major problems with edema (e.g., severe Cushing's syndrome, residual leg swelling from deep-vein thrombosis) No recent coronary artery disease No poorly controlled hypertension (diastolic greater than 110 mmHg and systolic greater than 180 mmHg) Pulmonary: DLCO greater than 80% of expected value Other: HIV negative No major psychiatric illness No other prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been free of disease for 5 years Not pregnant or nursing Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: No prior nitrosourea or temozolomide No more than 1 prior chemotherapy regimen allowed for patients with glioblastoma At least 6 weeks since mitomycin or procarbazine and recovered At least 4 weeks since other prior chemotherapy and recovered No other concurrent chemotherapy Endocrine therapy: If receiving steroids, must be on a stable steroid dose for at least 72 hours prior to study No other concurrent endocrine therapy Radiotherapy: At least 6 weeks since radiotherapy No greater than 10-20% of marrow irradiated in prior radiotherapy No other concurrent radiotherapy Surgery: Surgery allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82
Dates: Start 1998-03-25 (Actual); Primary Completion 2001-12-03 (Actual); Study Completion 2004-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Prados, MD, Study Chair — UCSF Medical Center at Parnassus
Locations (10):
- United States (10):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Chang SM, Prados MD, Yung WK, Fine H, Junck L, Greenberg H, Robins HI, Mehta M, Fink KL, Jaeckle KA, Kuhn J, Hess K, Schold C. Phase II study of neoadjuvant 1, 3-bis (2-chloroethyl)-1-nitrosourea and temozolomide for newly diagnosed anaplastic glioma: a North American Brain Tumor Consortium Trial. Cancer. 2004 Apr 15;100(8):1712-6. doi: 10.1002/cncr.20157. PMID 15073861
- [Result] Prados MD, Yung WK, Fine HA, Greenberg HS, Junck L, Chang SM, Nicholas MK, Robins HI, Mehta MP, Fink KL, Jaeckle KA, Kuhn J, Hess KR, Schold SC Jr; North American Brain Tumor Consortium study. Phase 2 study of BCNU and temozolomide for recurrent glioblastoma multiforme: North American Brain Tumor Consortium study. Neuro Oncol. 2004 Jan;6(1):33-7. doi: 10.1215/S1152851703000309. PMID 14769138